CLINICAL TRIAL: NCT06822803
Title: Effects of an Urban-gardening Nutrition Intervention for Food Insecure College Students
Acronym: UGNIFICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Principal Investigator, Catherine Coccia, PhD, RD, Associate Professor, Florida International University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-19-0134
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Food Insecurity; Obesity Prevention
Keywords: College student food insecurity; Gardening nutrition intervention; college students; nutrition education; social cognitive theory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gardening Nutrition Education Program (Experimental): Intervention group participants completed in person 1-hour educational sessions, once a week for 6 weeks, and completed the post test and anthropometric measurements on the 7th week. The sessions included nutrition education, recipes, cooking demos, home gardening tips, and a take home vertical garden. A satisfaction survey was also administered at the last educational session (week 6). Multiple weekly sessions were scheduled to accommodate the participants' schedules. Sessions were capped at 12 students to allow for a more personalized experience. Text messages were used weekly to remind the participants and confirm attendance for each session.
  Interventions: Behavioral: Gardening Nutrition Education Program
- Control Group (No Intervention): Participants in this group did not receive the intervention.

INTERVENTIONS:
Behavioral: Gardening Nutrition Education Program — This intervention was a 6-week Social Cognitive Theory based, urban gardening, cooking and nutrition education program designed to change health behavior mediators, fruit and vegetable intake, stress, and life satisfaction in food insecure college students.
  Arms: Gardening Nutrition Education Program

SUMMARY:
The goal of this clinical trial is to learn if an urban gardening nutrition education program can have positive health effects on food insecure college students. The main question it aims to answer is to determine whether an 8-week urban-gardening nutrition intervention can improve fruit and vegetable intake, nutrition knowledge, Body Mass Index (BMI) and body fat percentage in college students with food insecurity.

Participants will:

Fill out a questionnaire regarding demographics, food insecurity, fruit and vegetable intake, nutrition knowledge, self-efficacy and health beliefs.

Allow researchers to measure height, weight and body fat percentage Participate in a 1-hour education cooking or gardening session once a week for 8 weeks Receive text message reminders for meeting dates

ELIGIBILITY:
Inclusion Criteria:

* Must be enrolled at FIU
* Age 18+ years old
* Literate in English
* Food insecure

Exclusion Criteria:

* Students who are student athletes
* Women who are pregnant or planning to become pregnant in the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Mean Fruit and Vegetable Intake at 8 Weeks | From enrollment to the end of interventiont at 8 weeks
  Fruit and vegetable intake was measured using the National Cancer Institute's Fruit and Vegetable Screener as well as through a 1-item question, "Yesterday, how many servings of fruits and vegetables did you consume?" Higher numbers indicate higher levels of fruit and vegetable intake.
Change from Baseline in the Mean Stress Scores at 8 Weeks | From enrollment to the end of interventiont at 8 weeks
  Stress levels was measured using Cohen's Perceived Stress Scale. Higher numbers indicate higher levels of stress.
Change from Baseline in the Mean Life Satisfaction Scores at 8 Weeks | From enrollment to the end of interventiont at 8 weeks
  Life Satisfaction was measured using Diener's Quality of Life. Higher numbers indicate higher levels of life satisfaction.
Change from Baseline in the Mean Body Mass Index Scores at 8 Weeks | From enrollment to the end of interventiont at 8 weeks
  Anthropometrics were collected from all participants using standard techniques. Height was measured barefoot by stadiometer and weight was measured barefoot by a digital scale, with empty pockets and without heavy clothing such as sweaters. Participants will also self-report their height and weight for reference. BMI was calculated using the standard equation using height (cm) and weight (kg) Higher numbers indicate higher BMI.

SECONDARY OUTCOMES:
Change from Baseline in the Mean Nutrition Knowledge Scores | From enrollment to the end of intervention at 8 weeks
  Nutrition knowledge was measured using an adapted version of 20- item Dickson-Spillmann Consumer Oriented Nutrition Knowledge Survey (CoNKS). 10 population relevant True or False style questions were included. Higher numbers indicate higher levels of nutrition knowledge.
Change from Baseline in the Mean Self Efficacy, Outcome Expectation and Reciprocal Determinism | From enrollment to the end of intervention at 8 weeks
  Behavior change was measured through Social Cognitive Theory constructs. These will be measured through Dewar's SCT constructs scales. Higher numbers indicate higher levels of self-efficacy, outcome expectations and reciprocal determinism.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No